CLINICAL TRIAL: NCT02351128
Title: Traitement Des Carcinomes à Cellules de Merkel inopérables et/ou métastatiques Par Analogue de la Somatostatine - Etude Nationale Multicentrique Mono-bras de Phase II.
Brief Title: Treatment of Unresecable and/or Metastatic Merkel Cell Carcinoma by Somatostatine Analogues
Acronym: PHRC-Merkel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC14.040; 2014-001273-13 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Carcinoma, Merkel Cell
Keywords: lanreotide
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Only one arm (Experimental): All patients receive Lanreotide.
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide
  Other Names: Somatuline

SUMMARY:
The purpose of this trial is to evaluate the efficacy of lanreotide on locally evolving and/or metastatic MCC in a national prospective multicentre phase II study (centres belonging to the skin cancer task force of the French Society of Dermatology namely "Groupe de Cancérologie Cutanée de la Société Française de Dermatologie"). This one-arm study, for which the primary endpoint is overall response to lanreotide, will follow an A'Hern plan in one step (A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med 2001, 20:859-66) with main evaluation at 12 weeks on a population of 35 patients. The investigators make assumption that a 40% success rate at 3 months would be desirable, but if it was 20% or less the treatment would be unacceptable. It gives a trial size of 35 patients with a cut-off of 12 patients. Over 12 patients lanreotide will be considered as effective.

The lanreotide treatment (Somatuline LP 120 mg injected subcutaneously every 28 days) will be provided by IPSEN Pharma laboratory. An ancillary immunohistochemistry study on somatostatine receptors 2,3,5, dopamine receptors 1,2 and polyomavirus MCPyV will bring new data on this neuroendocrine tumour and potentially provide new therapeutic perspectives.

The results of this study may :

* determine whether somatostatin analogues may help to treat locally advanced and/or metastatic MCC;
* address whether there is a correlation between positive SPECT-CT (octreoscan) assessment and therapeutic response to lanreotide;
* evaluate the place of TEP-CT and SPECT-CT for MCC evaluation/staging;
* evaluate in future studies, with the ancillary data, other analogues or hybrid molecules;
* consider, if positive results are obtained from this study, somatostatin analogues as adjuvant treatment after surgery of primary MCC.

DETAILED DESCRIPTION:
The efficacy will be considered as success if patient have a positive response to lanreotide.

Primary criterion Positive response at 3 months will be defined according to the RECIST 1.1 criteria (clinical and TDM evaluation will be done at 3 months): complete response (CR) or partial response (PR) or stable disease (SD) at 3 months.

Secondary Objectives:

* Assessment of the primary criterion at M6, M9, M12, M18 and M24
* Description of the overall survival and time to progression
* Assessment of the efficacy of the following radiological exams for staging the disease: SPECT-CT and TEP-CT
* Description of the correlation of SPECT-CT results (positivity or negativity) and response to treatment, and the correlation of TEP-CT results and response to treatment
* Description of the safety and tolerability of lanreotide in this study

Population and Methods

Experimental plan French national prospective multicentre phase II one-arm study. This one-arm study, for which the primary endpoint is overall response to lanreotide, will follow an A'Hern plan in one step.

Population Inclusion criteria

* Histologically confirmed neuroendocrine carcinoma of the skin (Merkel cell carcinoma) with inoperable local-regional disease or distant metastatic disease (stages IIIB or IV AJCC 2010), cerebral nervous system metastases will be allowed.
* First line of treatment or more
* Measurable disease: at least 20 mm by conventional techniques or 10 mm by spiral CT scan
* Age 18 years or older;
* WHO performance status ECOG 0-3
* premenopausal patients must use effective contraception
* No other prior malignancy within 5 years except adequately treated basal cell or squamous cell carcinoma or in situ cancer of the cervix
* No other concurrent chemotherapy, immunotherapy or hormone therapy.
* At least 4 weeks since adjuvant chemotherapy, 14 days since radiotherapy and 2 weeks since surgery
* Biological functions: absolute neutrophil count at least 1000/mm3, platelet count at least 100000/mm3, haemoglobin at least 9g/dl (transfusion allowed), bilirubin no greater than 3 times upper limit of normal (ULN), SGOT and SGPT no greater than 2.5 times ULN, no untreated chronic liver disease, creatinine no greater than 1.5 times ULN, no untreated chronic renal disease, no untreated diabetes or infection
* Written informed consent

Exclusion criteria

* previous hypersensibility to lanreotide treatment
* complicated and untreated cholelithiasis
* pregnancy or breast-feeding
* patient treated with cyclosporine

Studied treatment Lanreotide 120 mg sub-cutaneously every 28 days during 12 weeks, followed by injections every 28 days if response is positive until progression. The expected rate of positive response is 50% of patients at 3 months and 25% of patients at 1 year.

Evaluation Criteria and follow-up of the study The inclusions will be done during 2 years and the follow-up of patients is planned to be 2 years, to have an optimal assessment of progression free survival in case of response to treatment, with a total study duration of 4 years.

Data collection

* at inclusion : patient's demography and medical history; clinical and anatomopathological data on primary MCC; blood count, platelets, electrolytes, glucose, creatinine, transaminases, bilirubin, ECG, pregnancy test for women of childbearing age;
* Clinical examination and measure of possible target lesions (tumor and cutaneous metastasis) using RECIST 1.1 criteria at inclusion and at M1, M2 and M3 and every 3 months during the first year (M6, M9 and M12) and every 6 months during the second year of follow-up (M18 and M24);
* Cerebral and thoraco-abdominal CTscan with results of imaging (RECIST 1.1 criteria: http://www.recist.com/recist-in-practice/01.html) at inclusion, at 3 months and, every 3 months during the first year, every 6 months during 2nd year;
* Octreoscan (SPECT-CT) at inclusion
* PET-CT at inclusion

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed neuroendocrine carcinoma of the skin (Merkel cell carcinoma) with inoperable local-regional disease or distant metastatic disease (stages IIIB or IV AJCC 2010), cerebral nervous system metastases will be allowed.
* First line of treatment or more
* Measurable disease: at least 20 mm by conventional techniques or 10 mm by spiral CT scan
* WHO performance status ECOG 0-3
* premenopausal patients must use effective contraception
* No other prior malignancy within 5 years except adequately treated basal cell or squamous cell carcinoma or in situ cancer of the cervix
* No other concurrent chemotherapy, immunotherapy or hormone therapy.
* At least 4 weeks since adjuvant chemotherapy, 14 days since radiotherapy and 2 weeks since surgery
* Biological functions: absolute neutrophil count at least 1000/mm3, platelet count at least 100000/mm3, haemoglobin at least 9g/dl (transfusion allowed), bilirubin no greater than 3 times upper limit of normal (ULN), SGOT and SGPT no greater than 2.5 times ULN, no untreated chronic liver disease, creatinine no greater than 1.5 times ULN, no untreated chronic renal disease, no untreated diabetes or infection
* Written informed consent

Exclusion Criteria:

* previous hypersensibility to lanreotide treatment
* complicated and untreated cholelithiasis
* pregnancy or breast-feeding
* patient treated with cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patient with positive response according to the RECIST 1.1 criteria | at 3 months
  Positive response will be defined according to the RECIST 1.1 criteria

SECONDARY OUTCOMES:
Percentage of patient with positive response according to the RECIST 1.1 criteria | at 6, 9,12,18 and 24 months
  Positive response will be defined according to the RECIST 1.1
Number of Participants with Adverse Events | at 3,6, 9,12,18 and 24 months
  Description of the safety and tolerability of lanreotide in this study

CONTACTS AND LOCATIONS:
Overall Officials: BEYLOT-BARY Marie, Principal Investigator — Bordeaux University Hospital, Haut-lévêque; DUTRIAUX Carole, Principal Investigator — Bordeaux University Hospital, St André; DALAC Sophie, Principal Investigator — Centre Hospitalier Universitaire Dijon; DUPUY Alain, Principal Investigator — Rennes University Hospital; LEBBE Céleste, Principal Investigator — AP-HP- Saint Louis; AVRIL Marie-Françoise, Principal Investigator — AP-HP - Cochin; DALLE Stéphane, Principal Investigator — HCL- Lyon Sud, Pierre Bénite; GUILLOT Bernard, Principal Investigator — Montpellier University Hospital; VERNEUIL Laurence, Principal Investigator — University Hospital, Caen; DRENO Brigitte, Principal Investigator — Nantes University Hospital; HAINAUT-Wierzbicka Ewa, Principal Investigator — Poitiers University Hospital; GROB Jean-Jacques, Principal Investigator — AP-HM; DEQUATREBARBES Julie, Principal Investigator — Annecy Interregional Hospital; ZEHOU Ouidad, Principal Investigator — AP-HP-Henri MONDOR
Locations (1):
- Grenoble University Hospital, Grenoble, France